CLINICAL TRIAL: NCT03850457
Title: The Incidence, Risk Factors, Diagnosis, Treatments and Burden of Bronchopulmonary Dysplasia (BPD) Among Very Preterm Infants in China: A Nationwide Prospective Cohort Study.
Brief Title: Epidemiological Study for Bronchopulmonary Dysplasia (BPD) in China
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shengjing Hospital (Other); Beijing Children's Hospital (Other); Inner Mongolia Maternity and Child Health Care Hospital (Unknown); Shanxi Provincial Maternity and Children's Hospital (Other); Qilu Children's Hospital of Shandong University (Other); The Affiliated Hospital of Qingdao University (Other); Yantai Yuhuangding Hospital (Other); Shanghai Children's Medical Center (Other); Shanghai First Maternal and Infant Health Hospital affiliated to Tongji University Medical School (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Nanjing Maternity and Child Health Care Hospital (Other); The First Affiliated Hospital of USTC (Unknown); Anhui Provincial Children's Hospital (Other); Yuying Children's Hospital of Wenzhou Medical College (Unknown); Ningbo Women & Children's Hospital (Other); QuanZhou Women and Children's Hospital (Other); Xiamen Maternity and Child Health Care Hospital (Unknown); The First Affiliated Hospital of Zhengzhou University (Other); Children's Hospital of Zhengzhou University (Unknown); Hubei Maternity and Child Health Care Hospital (Unknown); Hunan Children's Hospital (Other Government); Foshan Maternity and Child Health Care Hospital (Unknown); Maoming Maternity and Child Health Care Hospital (Unknown); Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other); Gansu Provincial Maternal and Child Health Care Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Xinjiang People's Hospital (Unknown); Chengdu Women and Children's Center Hospital (Other); Guizhou Maternity and Child Health Care Hospital (Unknown); The Affiliated Hospital of Zunyi Medical College (Unknown)
Responsible Party: Sponsor
Other Study IDs: EKYYBPDMC
Record Dates: First submitted 2019-01-28; First posted 2019-02-21 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: bronchopulmonary dysplasia; preterm infants; epidemiologic characteristics; risk factors; mortality
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — The treatments will be determined by their neonatologists and no additional investigational drugs will be applied to the infants included in this study.

SUMMARY:
This study will establish a nationwide cohort of very preterm infants in China, to investigate the epidemiological characteristics and short-term outcomes of BPD in different NICUs around the country.

DETAILED DESCRIPTION:
This is a nationwide multicenter prospective cohort study of very preterm infants in China. We will collect general information of very preterm infants, maternal and obstetrical conditions, resuscitation strategies in delivery room, diagnosis of BPD, treatments and complications from medical record review and family interviews.

This study aims to 1) investigate the epidemiologic characteristics of BPD based on the National Institutes of Health consensus definition in 2000 and 2016 respectively, and compare the applicability of two standard criteria for BPD in China; 2) identify independent risk factors for the development of BPD, such as ethnicity, gender, gestational age, birth weight, maternal and obstetrical conditions, fetal conditions, chorioamnionitis, infection, anemia, PDA, early pulmonary hypertension and so on; 3) establish prediction models of BPD at different postnatal ages; 4) investigate the short-term outcomes of BPD, such as mortality in NICU, LOS, late pulmonary hypertension, and so on; 5) investigate the prevention and treatment measures of BPD and evaluate the implementation of high evidence practices to reduce mortality and BPD, such as using antenatal steroids and caffeine; 6) investigate economic burden of BPD in China.

This program is organized by the steering committee, on which each clinical center and data coordinating center are represented. Each center will contribute to data collection and coordination. The steering committee will hold a conference call every month, meet in-person twice yearly and additionally hold working meetings at the Congress of Chinese Pediatric Society and the Congress of Chinese Neonatal Society. The committee will identify and resolve issues, encourage the centers to finish their work better. The data coordinating center will manage clinical report forms, provide support for standardization of definitions, data collection and quality control. The data coordinating center will hold training webinars with the research team from each site to ensure uniform approaches to data collection before study inception.

A centralized research electronic data capture system (by Suirong Corporation, Shanghai, China) will be used in this study. Each site will contribute data using a computer-based interface. Individual centers will retain access to their own data through customized downloads from the database management tool.

Data cleaning and statistical analysis will be conducted by an independent epidemiology & statistics work group from Children's Hospital of Fudan University and Public Health School of Fudan University. The study protocol and consent forms were evaluated by the institutional review board (IRB) of Fudan University. The protocol, questionnaire, statistical analysis plan and IRB approvals will be accessible on the website of China Neonatal Network.

ELIGIBILITY:
Inclusion Criteria:

* Infants with GA less than 32 weeks;
* Admitted to member neonatology centers during the period of recruitment;
* Age at admission less than 28 days.

Exclusion Criteria:

* Infants with major congenital anomalies, which include but not limited to serious congenital heart defects, chromosomal abnormalities, gastrointestinal atresias, brain malformations, congenital diaphragmatic hernia, renal agenesis or dysplastic kidneys;
* Infants with inborn errors of metabolism;
* Infants with severe heritable disease.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All neonates of gestational age less than 32 weeks
Sampling Method: Non-Probability Sample
Enrollment: 3800 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Bronchopulmonary dysplasia | 36 weeks of postmenstrual age
  Diagnosis by the standard criteria developed by NICHD in 2016 and 2000.
Mortality in NICU | through study completion, an average of 3 months
  The preterm infants who dies owing to persistent parenchymal lung disease or other diseases in NICUs.

SECONDARY OUTCOMES:
NICU length of stay (LOS) | through study completion, an average of 3 months
  The length of stay in NICU (days)
Hospital costs | through study completion, an average of 3 months
  The total costs in NICU (yuan)
Other complications | through study completion, an average of 1 year
  Such as NRDS, ROP, NEC, PDA, IVH, pneumothorax, pulmonary hypertension, pneumonia, apnea, hyperbilirubinemia, sepsis, anemia, CNS infection, and so on. All the complications will be diagnosed by the standard criteria made by China Neonatal Network.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Chen, MD,PhD, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ehrenkranz RA, Walsh MC, Vohr BR, Jobe AH, Wright LL, Fanaroff AA, Wrage LA, Poole K; National Institutes of Child Health and Human Development Neonatal Research Network. Validation of the National Institutes of Health consensus definition of bronchopulmonary dysplasia. Pediatrics. 2005 Dec;116(6):1353-60. doi: 10.1542/peds.2005-0249. PMID 16322158
- [Background] Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001 Jun;163(7):1723-9. doi: 10.1164/ajrccm.163.7.2011060. No abstract available. PMID 11401896
- [Background] Higgins RD, Jobe AH, Koso-Thomas M, Bancalari E, Viscardi RM, Hartert TV, Ryan RM, Kallapur SG, Steinhorn RH, Konduri GG, Davis SD, Thebaud B, Clyman RI, Collaco JM, Martin CR, Woods JC, Finer NN, Raju TNK. Bronchopulmonary Dysplasia: Executive Summary of a Workshop. J Pediatr. 2018 Jun;197:300-308. doi: 10.1016/j.jpeds.2018.01.043. Epub 2018 Mar 16. No abstract available. PMID 29551318
- [Background] Krishnan U, Feinstein JA, Adatia I, Austin ED, Mullen MP, Hopper RK, Hanna B, Romer L, Keller RL, Fineman J, Steinhorn R, Kinsella JP, Ivy DD, Rosenzweig EB, Raj U, Humpl T, Abman SH; Pediatric Pulmonary Hypertension Network (PPHNet). Evaluation and Management of Pulmonary Hypertension in Children with Bronchopulmonary Dysplasia. J Pediatr. 2017 Sep;188:24-34.e1. doi: 10.1016/j.jpeds.2017.05.029. Epub 2017 Jun 20. No abstract available. PMID 28645441
- [Derived] Dai Y, Sheng K, Hu L. Diagnostic efficacy of targeted high-throughput sequencing for lower respiratory infection in preterm infants. Am J Transl Res. 2022 Nov 15;14(11):8204-8214. eCollection 2022. PMID 36505277